CLINICAL TRIAL: NCT05201014
Title: CAncer Survivor CArdiomyopathy DEtection Pilot Study
Brief Title: Cancer Survivor Cardiomyopathy Detection
Acronym: CASCADE
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Florida Heart Research Institute (Other)
Responsible Party: Principal Investigator, Joerg Herrmann, MD, Professor of Medicine, Mayo Clinic
Other Study IDs: CASCADE; NCI-2022-05920 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); 21-006790 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-12-02; First posted 2022-01-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Cancer
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1 year follow-up: patients who were treated in the year before and are now returning for their 1-year follow-up.
  Interventions: Diagnostic Test: NT-pro-BNP; Diagnostic Test: Electrocardiogram; Diagnostic Test: Echocardiogram
- Prior to anthracycline-based therapy: patients presenting before the start of anthracycline-based therapy, then to be followed thereafter for 1 year and thereby contributing to the pool of patients with 1-year post-anthracycline assessment.
  Interventions: Diagnostic Test: NT-pro-BNP; Diagnostic Test: Electrocardiogram; Diagnostic Test: Echocardiogram

INTERVENTIONS:
Diagnostic Test: NT-pro-BNP — Blood draw
  Other Names: Blood Biomarker
Diagnostic Test: Electrocardiogram — electrodes are placed on certain spots and a reading obtained to measure the voltage of the heart
Diagnostic Test: Echocardiogram — medical imaging of the heart

SUMMARY:
The purpose of this study is to improve the cardiovascular care of adult cancer survivors. The goal is to obtain the data necessary to plan and develop a nation-wide network of a screening program that can help provide cost-effective and long-term monitoring.

DETAILED DESCRIPTION:
The primary objective of this study is to define the diagnostic performance and optimal cutoffs of AI-ECG and NT-pro-BNP for the detection of left ventricular dysfunction [LVD, defined as a left ventricular ejection fraction (LVEF) <50%] in cancer patients at 1 year after completion of anthracycline-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age prior to enrollment and anthracycline start date
* Diagnosis of breast cancer, lymphoma, or sarcoma with either planned or at 1 year after completion of anthracycline therapy, including patients from 6-12 months and greater than 1 year post-anthracycline exposure.
* Patients with a history of persistent atrial fibrillation (afib) that are not in afib remission. Include if the most recent ECG does not show afib. Atrial flutter treated the same

Exclusion Criteria:

* LVEF <50% or prior confirmed history of cardiomyopathy, heart failure, left bundle branch block, or paced rhythm
* Patients with a history of persistent atrial fibrillation (afib) that are not in afib remission. Include if the most recent ECG does not show afib. Atrial flutter treated the same.
* Individuals with pacemakers, defibrillators, or other implanted electronic devices
* Inability/unwillingness of individual to give written informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 cancer survivors who are 1 year out from anthracycline-based therapy.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of AI-ECG for left ventricular ejection fraction (LVEF) < 50% | 1 year post anthracycline therapy
  Determination of the sensitivity, specificity, positive and negative prediction value as well as area under the curve for receiver operating characteristics for the 12-lead AI ECG algorithm for an LVEF <50%
Diagnostic performance of NT-pro-BNP for left ventricular ejection fraction (LVEF) < 50% | 1 year post anthracycline therapy
  Determination of the sensitivity, specificity, positive and negative prediction value as well as area under the curve for receiver operating characteristics for NT-pro-BNP >125 for an LVEF <50%
Diagnostic performance of AI-ECG and NT-pro-BNP for left ventricular ejection fraction (LVEF) < 50% | 1 year post anthracycline therapy
  Determination of the sensitivity, specificity, positive and negative prediction value as well as area under the curve for receiver operating characteristics for the 12-lead AI ECG algorithm and NT-pro-BNP >125 combined for an LVEF <50%

SECONDARY OUTCOMES:
Absolute change in LVEF from baseline to 1 year from anthracycline-based therapy | 1 year
  Calculation of the the change in LVEF from baseline to 1 year from anthracycline-based therapy
Absolute change in AI-ECG probability for LVEF <50% from baseline to 1 year from anthracycline-based therapy | 1 year
  Calculation of the change in AI-ECG probability of LVEF <50% from baseline to 1 year from anthracycline-based therapy
Correlation of change in LVEF and AI-ECG probability of LVEF <50% from baseline to 1 year from anthracycline-based therapy | 1 year
  Calculation of the correlation coefficient of change in LVEF and AI-ECG probability of LVEF <50% from baseline to 1 year from anthracycline-based therapy
Absolute change in NT-pro-BNP from baseline to 1 year from anthracycline-based therapy | 1 year
  Calculation of the change NT-pro-BNP from baseline to 1 year from anthracycline-based therapy
Correlation of change in LVEF and NT-pro-BNP from baseline to 1 year from anthracycline-based therapy | 1 year
  Calculation of the correlation coefficient of change in LVEF and NT-pro-BNP from baseline to 1 year from anthracycline-based therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Herrmann, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials